CLINICAL TRIAL: NCT03987893
Title: Therapeutic Efficacy of Oral PEG3350 Plus Lactulose Versus Lactulose Alone in Patients of Acute on Chronic Liver Failure With Overt Hepatic Encephalopathy: A Single Blind Prospective Randomized Controlled Study
Brief Title: PEG3350 in ACLF With Hepatic Encephalopathy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Radha K Dhiman, Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT/IEC/2018-000485
Record Dates: First submitted 2019-06-13; First posted 2019-06-17 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Hepatic Encephalopathy; Acute-On-Chronic Liver Failure
Keywords: PEG3350; hepatic encephalopathy; acute on chronic liver failure; lactulose; rifaximin; HESA
MeSH Terms: conditions — Hepatic Encephalopathy; Acute-On-Chronic Liver Failure | interventions — polyethylene glycol 3350; Lactulose

STUDY DESIGN:
Intervention Model Description: Open Label, randomized control trial
Masking Description: participant is randomised using a table of random numbers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PEG+Lactulose (Experimental): this arm will recieve PEG3350 in addition to standard of care
  Interventions: Drug: PEG-3350 with Electolytes; Drug: Lactulose
- Lactulose alone (Active Comparator): this arm will recieve only standard of care for management of hepatic encephlaopathy with ACLF
  Interventions: Drug: Lactulose

INTERVENTIONS:
Drug: PEG-3350 with Electolytes — experimental arm will receive 2 doses of PEG3350 spaced over 12 hours after randomization to arm1. PEG as dose of 2litres (1 sachet dissolved in 2L of water) will be administered via a nasogastric tube.
  Arms: PEG+Lactulose
Drug: Lactulose — Lactulose will be given orally (30ml QID) which shall be titrated to ensure 2-3 soft stools per day
  Other Names: Lactulose per orally

SUMMARY:
it is a single blind randomised control study which aims to study the effect of PEG3350 in resolution of overt hepatic encephalopathy in patients of acute on chronic liver failure. this will be compared with the standard of care in the management of hepatic encephalopathy.

DETAILED DESCRIPTION:
Therapeutic Efficacy of oral PEG3350 plus Lactulose Versus Lactulose alone in Patients of Acute on Chronic Liver Failure with Overt Hepatic Encephalopathy: A Single Blind Prospective Randomized Controlled Study

INTRODUCTION:

Hepatic encephalopathy (HE) refers to syndrome observed in patients with cirrhosis exhibiting clinical manifestations of mild to severe cognitive dysfunction (neuropsychiatric abnormalities) characterised by alterations in sleep pattern, sudden behavioural changes & personality changes along with altered cognition, or coma. The basic pathophysiology involved in development of potentially reversible neuropsychiatric abnormalities associated with HE are not clearly understood but ammonia generation by gut microbiota is considered as significant contributing factor. HE is categorized into overt hepatic encephalopathy (OHE) and minimal hepatic encephalopathy (MHE). Previous studies have reported the incidence of OHE and MHE to be 30-45% and 60-80% respectively in patients suffering from cirrhosis .

In the present study, we propose to assess the efficacy of an ammonia reducing therapy utilisisng PEG 3350 in patients with Acute on Chronic Liver Failure (ACLF).

Hepatic encephalopathy in Acute on Chronic Liver Failure (ACLF) The syndrome of acute on chronic liver failure is a recently described clinical entity. The defining criterion for acute-on-chronic liver failure (ACLF) takes into consideration the existence of hepatic encephalopathy (HE) within 4 weeks. In Asia, the following definition has been suggested: "acute hepatic insult manifesting as jaundice (serum bilirubin level ≥5 mg/dl) and coagulopathy (international normalized ratio ≥1.5), complicated within 4 weeks by ascites and/or encephalopathy in a patient with previously diagnosed or undiagnosed chronic liver disease" . In the West, experts proposed to define ACLF as "an acute deterioration of liver function in patients with cirrhosis which is usually associated with a precipitating event and results in the failure of one or more organs and high short-term mortality". This definition is on the basis of the European Association for the Study of the Liver (EASL)-Chronic Liver Failure (CLIF) Consortium Acute-on-Chronic Liver Failure in Cirrhosis (CANONIC)" study which established diagnostic criteria for ACLF in hospitalized patients who had an acute decompensation (AD) of cirrhosis . In ACLF, hyperammonemia, systemic inflammatory state mediated by various cytokines which includes sepsis/SIRS, bacterial translocation, insulin resistance resulting in hyperglycemia and oxidant induced injury, in addition modulation by glutaminase gene alteration along with alterations in cerebral hemodynamics appear to be crucial factors in the pathogenesis of encephalopathy.Various studies have explored the potential of bacterial infections, hyponatremia, alcohol intake and factors responsible for systemic inflammation in HE. HE is diagnosed after excluding other causes of altered cognition such as metabolic, neurological and psychiatric conditions. Clinical features of HE in ACLF patients are very much similar to those with HE in acute liver failure (ALF). The clear correlation of serum ammonia levels, systemic inflammation and outcome of HE in ACLF patients is not well understood .

Factors precipitating, HE, such as constipation, hyponatremia, infections etc. must be promptly identified and addressed appropriately. Currently Evidence-based medicine approach for the management of HE is restricted to early bowel evacuation and administration of non-absorbable antibiotics such as rifaximin. Antibiotics, prebiotics, treatment of diabetes and other supportive management reduces the systemic inflammation .

Most of the therapy regimens in treatment of hepatic encephalopathy are directed towards reduction of the generation of nitrogenous products, for which gut is the major site of generation and the organ of accumulation of nitrogenous toxins especially Ammonia in patients with liver failure and portosystemic shunting Treatment of Hepatic Encephalopathy Lactulose (beta-1,4-galactosido-fructose) has been used in practice for the management of HE because of its ammonia lowering effects . The mechanism by which lactulose act still remains controversial and is hypothesized to be by following methods, first is metabolism of lactulose by gut bacteria release organic acids which play vital role in trapping ammonium ions, second is by elimination of ammonia generating organisms and third is by replacing amminogenic organisms with urease lacking acidophilic bacteria . The role of inhibition of glutamine followed by decreased ammonia genesis has also been considered. Management and treatment of patients with OHE is mainly focused on elimination of underlying precipitating factors, nutritional supports, and lowering ammonemia . Lactulose and rifaximin are the most widely used medications to lower ammonia generation; however, their exact mechanism of action is still not well understood .

REVIEW OF LITERATURE:

Proposed Role of PEG 3350 in HE Before the routine use of non-absorbable disaccharides, simple laxatives were used in the management of hepatic encephalopathy assuming the beneficial effects of bowel evacuation in resolution of neurocognitive disturbances in liver diseases. With this principle, there were trials done assessing the clinical benefits of PEG solution, which is a commonly used laxative is used routinely in bowel preparation for colonoscopy. Currently there is a significant data showing the beneficial effects of PEG 3350 in overt HE due to underlying cirrhosis, however its efficacy in ACLF remains to be looked into. Similar to lactulose, polyethylene glycol is unabsorbed from the gut but in addition it also lacks the unabsorbed carbohydrate load which aids in lowering of stool pH and enhancing the amount of water lost from the stools. Furthermore, the rate of ammonia excretion via feces is enhanced with PEG as compared to lactulose. In this study, we propose to evaluate the efficacy & safety profile of PEG3350 plus lactulose vs. lactulose alone for treatment of ACLF. An essential understanding required with PEG usage is to consider that it exerts a significant cathartic effect and thus may progress to dehydration, hypovolemia, dyselectrolemia, and even blood gas abnormalities. It's also the most prominently used preparative agent in patients undergoing colonoscopy, and is thus widely used in human population worldwide. PEG preparations are easily available and are cost effective. Another potential benefit of utilizing PEG for OHE is that it may result in decrease in the duration of hospitalization, depending on the causes of the HE. By accelerating the treatment of hepatic encephalopathy, PEG can help patients to return to normal life more rapidly and decrease the direct and indirect cost of illness caused by hepatic encephalopathy. PEG, which resolves decreased level of consciousness more effectively and more rapidly in the first 24 hours, can also help physicians to identify the other causes of altered mental status more quickly and more accurately.

Some of the trials which have compared the efficacy of PEG in management of HE are:

Author Trial Conclusion. Rahimi et al., (n=50) "Lactulose vs Polyethylene Glycol 3350-Electrolyte Solution for Treatment of Overt Hepatic Encephalopathy The HELP Randomized Clinical Trial" "PEG led to more rapid HE resolution than standard therapy".

Naderian et al., (n=40) "Polyethylene Glycol and Lactulose versus Lactulose Alone in the Treatment of Hepatic Encephalopathy in Patients with Cirrhosis: A Non-Inferiority Randomized Controlled Trial" "The use of PEG along with lactulose in comparison with lactulose alone is more effective in the treatment of hepatic encephalopathy in patients with cir¬rhosis".

Patients and methods:

Study Design: A prospective interventional cohort study using the drug PEG3350 + lactulose versus lactulose alone.

Allocation: randomized Intervention model: parallel assignment Masking: none, open label Primary purpose: treatment. Setting: Academic hospital - PGI (Chandigarh, India). Patients fulfilling eligibility criteria will be approached for informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years.
* Patients with ACLF with presence of hepatic encephalopathy > grade 2 as per WHC

Exclusion Criteria:

* Pregnant women or those who are suspected to be having acute fatty liver of pregnancy
* Malarial hepatopathy, enteric hepatitis, or ischemic hepatitis.
* Serum Na <125 mEq/litre
* Gastrointestinal (GI) obstruction, ileus, or gastric retention
* Bowel perforation
* Toxic colitis or toxic megacolon
* Structural brain lesions (as indicated by computed tomography imaging if available and confirmed by neurological exam)
* Other causes of altered mental status (i.e. not meeting the definition of hepatic encephalopathy
* Uncontrolled infection with hemodynamic instability requiring vasopressors.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-20 (Actual); Primary Completion 2020-05-25 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
Improvement in survival. | At day 28 and day 90.
  to look for any survival benefit in experimental arm at 28 days and 90 days
Improvement of encephalopathy by one or more grades. | 24 hours, 48 hours and 72 hours
  to look for the degree of improvement in grade of HE in both experimental arm and lactulose arm.

SECONDARY OUTCOMES:
Reduction in ammonia levels during and at the end of 48 hours, 72 hours and lactulose administration | 24 hours, 48 hours and 72 hours
  to extrapolate weather reduction of grade of HE correlates with reduction of ammonia levels
Prolongation of time to death among non-survivors. | 30 days
  to analyse the difference in time to event(death) among non survivors in experimental arm
Prevention / reduction of cerebral edema | 72 hours
  to look for any evidence of cerebral edema reduction by means of optic nerve sheath diameter
Reduction of seizures frequency | 30 days
  to analyse if reduction of HEresults in reduction or prevention of seizure episodes in both arms

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Premkumar, DM, Study Chair — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate Institute of Medical Education and Research, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ahmed S, Premkumar M, Dhiman RK, Kulkarni AV, Imran R, Duseja A, Kaur P, Taneja S, Singh V, Mishra S, Roy A, Mehtani R. Combined PEG3350 Plus Lactulose Results in Early Resolution of Hepatic Encephalopathy and Improved 28-Day Survival in Acute-on-Chronic Liver Failure. J Clin Gastroenterol. 2022 Jan 1;56(1):e11-e19. doi: 10.1097/MCG.0000000000001450. PMID 33060437